CLINICAL TRIAL: NCT00087555
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Trial Comparing the Effects of Orally Administered Xyrem(R) (Sodium Oxybate) With Placebo for the Treatment of Fibromyalgia
Brief Title: Trial Comparing the Effects of Xyrem (Sodium Oxybate) With Placebo for the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Senior Director Clinical Development, Jazz Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMC-SXB-26
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2012-01-10 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Sodium Oxybate; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Experimental): Sodium oxybate 6.0 g per day.
  Interventions: Drug: Xyrem (sodium oxybate) oral solution
- 3 (Placebo Comparator): Placebo (one of two doses matching active treatment by volume).
  Interventions: Drug: Placebo
- 1 (Experimental): Sodium oxybate 4.5 g per day.
  Interventions: Drug: Xyrem (sodium oxybate) oral solution

INTERVENTIONS:
Drug: Xyrem (sodium oxybate) oral solution — Xyrem (sodium oxybate) oral solution 4.5 g per day in divided doses, 2.25 g at bedtime and another 2.5 g two and a half to four hours later for 8 weeks.
  Arms: 1
Drug: Xyrem (sodium oxybate) oral solution — Xyrem (sodium oxybate) oral solution 6.0 g per night in divided doses of 3 g at bedtime and 3 g at 2.5 to 4 hours later for 8 weeks.
  Arms: 2
Drug: Placebo — Placebo one of two doses matching active treatment by volume for 8 weeks.
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether Xyrem (sodium oxybate) is effective when used alone to treat the pain and sleep disturbances of fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia affects millions of Americans, yet there are no FDA approved drugs to treat this debilitating condition. Besides causing pain, it also disrupts normal sleep patterns in many of its victims. Pain and lack of sleep reinforce each other, making patients progressively more miserable. Xyrem is a potent hypnotic that induces and consolidates sleep. In a few small studies Xyrem has been reported to offer relief to some fibromyalgia patients. This trial is designed to test this hypothesis. Patients who enroll in this study will stop taking any prescription medications for fibromyalgia (over-the-counter pain relievers will be permitted). They will then take either Xyrem alone or placebo alone. Patients will be followed for eight weeks to evaluate any relief of the pain or functional impairment of fibromyalgia from their study treatment. Sleep characteristics will also be assessed subjectively and by polysomnographic recordings at baseline and twice during the treatment phase.

ELIGIBILITY:
Inclusion Criteria

* Sign & date informed consent
* Willing & able to complete trial as described in protocol
* > 18 years of age
* Meet American College of Rheumatology criteria for Fibromyalgia [Widespread pain for at least 3 months, including all of the following: (1) Pain on right & left sides of body; (2) Pain above & below waist; (3) Pain in axial skeleton; 4) Pain on digital palpation with approximately 4kg force in at least 11 of 18 tender point sites]
* (Study continuation) Have an average VAS pain score > 4 on a scale of 0 to 10 as recorded in patient diary the last week before Visit 4.
* Discontinue all prescription medication taken for fibromyalgia, including opiates, benzodiazepines, anticonvulsants taken for pain, antidepressants, cyclobenzaprine (Flexeril), and/or tramadol (Ultram) until study completion
* Continue all pre-existing nutritional and/or exercise regimens and/or behavioral, massage, acupuncture, physical or cognitive therapies on an unchanged, consistent & regular schedule throughout study
* Use only acetaminophen or over-the-counter non-steroidal anti-inflammatory drugs as rescue pain medications & to limit dose to the labeled over-the-counter maximum. Aspirin may only be used as a cardiac protectant; formulations with caffeine are excluded.
* Forego ingestion of alcohol for duration of study.
* Fertile females must use a medically accepted method of birth control (e.g., barrier method with spermicide, oral contraceptive, or abstinence) for duration of trial.

Exclusion Criteria

1. Have any of the following medical conditions:

   * Other rheumatic disease, such as rheumatoid arthritis, osteoarthritis, or systemic lupus erythematosis
   * Uncontrolled hypo- or hyper-thyroidism of any type
   * Unstable cardiovascular, endocrine, neoplastic (excluding localized basal cell carcinoma), gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurological, pulmonary, and/or renal disease which would place patient at risk during trial or compromise objectives outlined in protocol
   * Myocardial infarction within last six months
   * On their screening PSG (polysomnogram) have an Apnea Index greater than 10 per hour or an Apnea Hypopnea Index greater than 15 per hour. Note: patients with sleep apnea are not excluded if their indices are below these thresholds while sleeping with CPAP (Continuous Positive Airway Pressure) and they are compliant with CPAP therapy.
   * Problems that, in the investigator's opinion, would preclude the patient's participation and completion of this trial or compromise reliable representation of subjective symptoms.
   * If a patient will have to discontinue antidepressant medication taken for depression, the investigator must make an evaluation as to any risks from cessation of anti-depressant therapy. If, in the opinion of the investigator, a reasonable risk of resultant patient harm exists, patient is excluded from study participation
   * Current or recent history of substance abuse including alcohol abuse
   * History of seizure disorder, history of head trauma, migraine headaches or intracranial surgery, & are taking anticonvulsants
   * Succinic semialdehyde dehydrogenase deficiency
2. Have taken any of these therapies:

   * gamma-hydroxybutyrate (sodium oxybate) in 30 days prior to signing informed consent
   * any investigational therapy in 30 days prior to signing informed consent
   * ever taken anticonvulsants to treat epilepsy or any other convulsions
3. Unwilling to stop these therapies during course of trial:

   * anticonvulsants prescribed solely for pain
   * all antidepressants
   * medication for sleep
4. Have any of the following clinical laboratory results:

   * Serum creatinine > 2.0 mg/dL
   * TSH (Thyroid Stimulating Hormone) < 0.3 μU/mL OR TSH > 6 μU/mL
   * abnormal liver function tests (SGOT [AST] or SGPT [ALT] more than twice the upper limit of normal)
   * elevated serum bilirubin (more than 1.5 times the upper limit of normal)
   * pre-trial ECG with arrhythmia, greater than a first degree AV block
   * positive pregnancy test at any time during trial
5. Have any of the following socio-economic factors:

   * Pending worker's compensation litigation or related other monetary settlements
   * Have an occupation that requires variable shift work or routine night shifts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2004-07; Primary Completion 2005-04 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Zheng, MD, Study Director — Jazz Pharmaceuticals, Inc
Locations (20):
- United States (20):
  - Radiant Research, Scottsdale, Arizona
  - Osteoporosis Medical Center, Beverly Hills, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Miami Research Associates, Miami, Florida
  - Radiant Research, Inc., West Palm Beach, Florida
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Richard N. Podell, MD, Springfield, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Alvin Daughtridge Arthritis Center, Lenoir, North Carolina
  - C.A.R.E. Center, Raleigh, North Carolina
  - Cleveland Sleep Center, Middlebrook Heights, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Abigail Rebecca Neiman, MD, Katy, Texas
  - The University of Texas Health Science Center, San Antonio, Texas
  - Stress Medicine Clinic -- HealthSouth Rehabilitation Hospital, Sandy City, Utah
  - Pacific Rheumatology Research, Inc., Renton, Washington
  - Seattle Rheumatology Associates, Seattle, Washington

REFERENCES:
- [Background] A randomized, double blind, placebo-controlled multicenter trial comparing the effects of three doses of orally administered sodium oxybate with placebo for the treatment of narcolepsy. Sleep. 2002 Feb 1;25(1):42-9. PMID 11833860
- [Background] A 12-month, open-label, multicenter extension trial of orally administered sodium oxybate for the treatment of narcolepsy. Sleep. 2003 Feb 1;26(1):31-5. PMID 12627729
- [Background] U.S. Xyrem Multicenter Study Group. Sodium oxybate demonstrates long-term efficacy for the treatment of cataplexy in patients with narcolepsy. Sleep Med. 2004 Mar;5(2):119-23. doi: 10.1016/j.sleep.2003.11.002. PMID 15033130
- [Background] The abrupt cessation of therapeutically administered sodium oxybate (GHB) does not cause withdrawal symptoms. J Toxicol Clin Toxicol. 2003;41(2):131-5. doi: 10.1081/clt-120019128. PMID 12733850
- [Background] Scharf MB, Baumann M, Berkowitz DV. The effects of sodium oxybate on clinical symptoms and sleep patterns in patients with fibromyalgia. J Rheumatol. 2003 May;30(5):1070-4. PMID 12734908
- [Background] Russell IJ, Perkins AT, Michalek JE; Oxybate SXB-26 Fibromyalgia Syndrome Study Group. Sodium oxybate relieves pain and improves function in fibromyalgia syndrome: a randomized, double-blind, placebo-controlled, multicenter clinical trial. Arthritis Rheum. 2009 Jan;60(1):299-309. doi: 10.1002/art.24142. PMID 19116896

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo taken as two equally divided nightly doses
- Xyrem (Sodium Oxybate) 4.5g: Xyrem 4.5g taken as two equally divided nightly doses
- Xyrem (Sodium Oxybate) 6.0g: Xyrem 6.0g taken as two equally divided nightly doses
Period: Overall Study
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g
Started | 66 | 62 | 67
Treated | 65 | 60 | 67
Completed | 54 | 51 | 46
Not Completed | 12 | 11 | 21
Not completed — Adverse Event | 3 | 6 | 14
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Non - Compliance | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Screen Failure | 1 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Non Compliance | 0 | 0 | 1
Not completed — Chronic Migraine Headaches (Med History) | 1 | 0 | 0
Not completed — Patient wanted to go back on Med | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g | Total
Number analyzed (Participants) | 66 | 62 | 67 | 195
Age Continuous [Mean (Standard Deviation); unit: years] | 47.2 (10.69) | 47.2 (11.89) | 45.1 (11.51) | 46.5 (11.35)
Age, Customized [Number; unit: participants]
  18 - 39 Years | 16 | 14 | 23 | 53
  40 - 49 Years | 24 | 19 | 17 | 60
  50 - 64 Years | 22 | 26 | 25 | 73
  >=65 years | 4 | 3 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 58 | 64 | 184
  Male | 4 | 4 | 3 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 59 | 56 | 65 | 180
  African American | 4 | 6 | 1 | 11
  Asian | 0 | 0 | 1 | 1
  Hispanic | 2 | 0 | 0 | 2
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 66 | 62 | 67 | 195

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was a Composite of Changes From Baseline in Three Co-primary Self Report Measures: Pain Visual Analog Scale (PVAS, Electronic Diaries), Fibromyalgia Impact Questionnaire (FIQ), and Patient Global Impression of Change (PGI-C).
Description: The percentage of participants who met all 3 of the following criteria:
  Reduction of >=20% from baseline to week 8 in both PVAS & FIQ total score and PGI-C response of "very much better" or "much better". Analysis was based on LOCF (Last Observation Carried Forward) data. The PVAS ranges from 0 (no pain) to 100 (worst imaginable pain). The FIQ ranges from 0 (best function) to 100 (worst function). PGI-C is a 7 point likert scale measuring change in the participant's fibromyalgia symptoms that ranges from "very much worse" to "very much better"
Time Frame: Baseline to week 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g
Number analyzed (Participants) | 66 | 62 | 67
Percentage of Participants
  Responders | 12.9 | 29.8 | 28.1
  Non - Responders | 87.1 | 70.2 | 71.9
Statistical Analysis 1: Comparison: Placebo vs Xyrem (Sodium Oxybate) 4.5g vs Xyrem (Sodium Oxybate) 6.0g; Test type: Superiority or Other; p = 0.052, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Xyrem (Sodium Oxybate) 4.5g; Test type: Superiority or Other; p = 0.024, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Xyrem (Sodium Oxybate) 6.0g; Test type: Superiority or Other; p = 0.035, Chi-squared

ADVERSE EVENTS:
Arm/Group | Placebo | Xyrem (Sodium Oxybate) 4.5g | Xyrem (Sodium Oxybate) 6.0g
Serious Adverse Events (participants affected / at risk) | 0/65 | 1/60 | 1/67
Other Adverse Events (participants affected / at risk) | 39/65 | 41/60 | 52/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Xyrem (Sodium Oxybate) 4.5g (N=60) | Xyrem (Sodium Oxybate) 6.0g (N=67)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Xyrem (Sodium Oxybate) 4.5g (N=60) | Xyrem (Sodium Oxybate) 6.0g (N=67)
Nausea (Gastrointestinal disorders) | 6 | 10 | 19
Vomiting (Gastrointestinal disorders) | 0 | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 9
Sinusitis (Infections and infestations) | 2 | 3 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Headache (Nervous system disorders) | 4 | 8 | 11
Dizziness (Nervous system disorders) | 2 | 5 | 12
Paraesthesia (Nervous system disorders) | 1 | 4 | 1
Insomnia (Psychiatric disorders) | 1 | 4 | 2
Anxiety (Psychiatric disorders) | 0 | 3 | 1
Restlessness (Psychiatric disorders) | 0 | 3 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 4
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Eye Irritation (Eye disorders) | 1 | 1 | 0
Mydriasis (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 0 | 0
Abdominal Pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 2
Oedema Peripheral (General disorders) | 1 | 1 | 2
Irritability (General disorders) | 0 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 1
Feeling Hot (General disorders) | 0 | 0 | 2
Hangover (General disorders) | 0 | 0 | 2
Influenza Like Illness (General disorders) | 1 | 0 | 1
Thirst Decreased (General disorders) | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1
Feeling Drunk (General disorders) | 0 | 0 | 1
Feeling Jittery (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 2 | 2
Viral Infection (Infections and infestations) | 1 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 2
Cystitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 2 | 0 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Calcium Increased (Investigations) | 1 | 0 | 0
Heart Rate Increased (Investigations) | 1 | 0 | 0
Heart Rate Irregular (Investigations) | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 1 | 0
Weight Increased (Investigations) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Increased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes Mellitus Insulin-Dependent (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 3
Migraine (Nervous system disorders) | 0 | 1 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 2
Akathisia (Nervous system disorders) | 0 | 1 | 0
Balance Disorder (Nervous system disorders) | 0 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 1
Paralysis (Nervous system disorders) | 0 | 0 | 1
Sedation (Nervous system disorders) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 2 | 2
Abnormal Dreams (Psychiatric disorders) | 2 | 2 | 0
Agitation (Psychiatric disorders) | 1 | 2 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 2
Nightmare (Psychiatric disorders) | 0 | 0 | 2
Affect Lability (Psychiatric disorders) | 1 | 0 | 0
Anger (Psychiatric disorders) | 1 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 1
Bipolar Disorder (Psychiatric disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 0 | 1
Emotional Disorder (Psychiatric disorders) | 0 | 0 | 1
Frustration (Psychiatric disorders) | 0 | 0 | 1
Initial Insomnia (Psychiatric disorders) | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Panic Attack (Psychiatric disorders) | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0
Sleep Walking (Psychiatric disorders) | 0 | 0 | 1
Thinking Abnormal (Psychiatric disorders) | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 1
Urine Odour Abnormal (Renal and urinary disorders) | 0 | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2
Hot Flush (Vascular disorders) | 0 | 2 | 0
Poor Peripheral Circulation (Vascular disorders) | 1 | 0 | 0
Raynaud's Phenomenon (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other